CLINICAL TRIAL: NCT02810613
Title: Leiden University Medical Center Mini Donor Bank
Status: Withdrawn | Type: Observational
Why Stopped: Study never started.
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Meta Roestenberg, MD, PhD, Leiden University Medical Center
Other Study IDs: Mini Donor Bank
Record Dates: First submitted 2016-05-31; First posted 2016-06-23 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Malaria; Schistosoma Mansoni; Schistosoma Haematobium; Diabetes; Asthma
MeSH Terms: conditions — Malaria; Schistosomiasis; Schistosomiasis haematobia; Diabetes Mellitus; Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: No

SUMMARY:
(Bio)medical research, particularly immunological, metabolic, transcriptional or biological assays, occasionally require the use of fresh blood (peripheral mononuclear cells) or urine. In order to comply with international guidelines for Good Clinical Practice, the investigators propose to establish a Mini Donor Bank to be able to obtain fresh blood or urine from voluntary donors. Recruitment of volunteers will be a continuous process. Volunteers will consent to occasional blood- or urine donation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged ≥ 18 and ≤ 65 years and in good health.
2. Subject has adequate understanding of the procedures of the study.
3. Subject is able to communicate well with the investigator.
4. Subject has signed informed consent.
5. Subject refrains from donation to the Sanquin blood bank.

Exclusion Criteria:

1. Previous vasovagal collapse during venepuncture.
2. For female participants: pregnancy or lactation.
3. Presence of any chronic systemic condition, which could compromise the health of the volunteer when performing venepuncture or interfere with the interpretation of immunological or metabolic test results.
4. Chronic use of immunosuppressive drugs.
5. Total blood volume donated exceeding >500 mL in the past 4 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy human volunteers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
A collection of samples for the purpose of (bio)medical laboratory assays including immunological, metabolic, transcriptional or biological analyses. | 10 years
  collection of samples for the purpose of biomedical assays, e.g. biobanking of samples for different assays, each one of which has a separate objective

IPD SHARING:
Plan to Share IPD: No